CLINICAL TRIAL: NCT07225764
Title: Empiric vs Selective Medical Therapy for Calcium Oxalate Stone Prevention: A Randomized Controlled Trial
Brief Title: CaOx Stone Prevention
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mantu Gupta, Chair of Urology, MSW and MSM Hospitals Professor, Icahn School of Medicine at Mount Sinai Director of Endourology, Mount Sinai Medical Center, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY-25-00784
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Kidney Stones
Keywords: kidney stones; calcium oxalate; nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis | interventions — Chlorthalidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empiric Therapy (Experimental): Patients randomized to the empiric group will receive treatment based on the pH on urinalysis and stone composition. Patients with greater than 50% calcium oxalate monohydrate (COM) stone composition will be counseled on a low oxalate diet by a medical provider. Patients with greater than 50% calcium oxalate dihydrate (COD) stone composition will be prescribed 25 mg of chlorthalidone once a day. In the rare event the stone composition is 50% COM and 50% COD, then those patients will receive both low oxalate diet counseling and a prescription for chlorthalidone.
  Interventions: Drug: Chlorthalidone; Behavioral: Low oxalate diet
- Selective Therapy (Active Comparator): Patients randomized to the selective group will undergo medical therapy based on the American Urological Association (AUA) guidelines from the 24-hour urine collection results. Patients with idiopathic hyperoxaluria (> 40mg/day) will receive a low oxalate diet and receive the same dietary counseling, handout, and questionnaire as the empiric group. Patients with idiopathic hypercalciuria (> 250mg in men, >200mg in women) will be prescribed 25mg of chlorthalidone once a day.
  Interventions: Drug: Chlorthalidone; Behavioral: Low oxalate diet

INTERVENTIONS:
Drug: Chlorthalidone — Chlorthalidone 25 mg orally once daily is used to reduce urinary calcium excretion and prevent recurrent calcium-containing kidney stones. In this study, it is prescribed either based on stone composition (empiric group) or guided by 24-hour urine results (selective group) for participants meeting criteria for hypercalciuria or calcium oxalate dihydrate stones.
Behavioral: Low oxalate diet — Participants receive counseling to follow a low oxalate diet, limiting high oxalate foods (>50 mg/100 g) and restricting moderate oxalate foods (<50 mg/100 g) to a single four-ounce serving per day. The diet is prescribed either based on stone composition (empiric group) or guided by 24-hour urine results (selective group) for participants with idiopathic hyperoxaluria or calcium oxalate monohydrate stones.

SUMMARY:
This single-center randomized controlled trial at Mount Sinai West will enroll 80 patients undergoing percutaneous nephrolithotomy for calcium oxalate stones. Participants will be randomized to receive either empiric therapy or selective therapy guided by 24-hour urine evaluation. The primary outcome is change in calcium oxalate supersaturation at 4 weeks, aiming to determine whether empiric therapy can provide outcomes comparable to selective therapy while simplifying access to prevention.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled trial evaluating the effectiveness of empiric versus selective medical therapy for the prevention of calcium oxalate kidney stones. The study will enroll 80 patients at Mount Sinai West undergoing percutaneous nephrolithotomy (PCNL) for predominantly calcium oxalate stones. Participants will be randomized postoperatively to receive either empiric therapy (based on stone composition and urinalysis) or selective therapy (based on 24-hour urine metabolic evaluation). The primary endpoint is the change in calcium oxalate supersaturation (ssCaOx) at 4 weeks post-treatment. The study is designed to determine whether an empiric approach can achieve comparable outcomes to selective therapy while simplifying access to preventive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult age of 18 years
* Diagnosed with kidney stones and scheduled for PCNL.
* Calcium Oxalate Stone Former
* Pre-operative CT-scan within 90 days of surgery and stone density with > 1000 Hounsfield units
* Non-pregnant or breastfeeding
* Able and willing to provide informed consent.
* Pre-operative eGFR greater than 70 mL/min/1.73 m² -Negative pre-operative urine culture

Exclusion Criteria:

* Documented history of gastric or intestinal bypass, liver disease, history of gastrointestinal malabsorptive disease (Crohn's disease, ulcerative colitis, and short-gut syndrome)
* Hyperparathyroidism -Renal tubular acidosis
* Active kidney stone prevention treatment (use of thiazides, alkaline therapy, or low oxalate diet) at the time of surgery
* History of hypokalemia or baseline hypotension
* Allergy to medications used in trial or sulfa-containing medications
* Patient prescribed thiazide, loop diuretics, carbonic anhydrase inhibitors, xanthine oxidase inhibitors, active Vitamin D, bisphosphonates, denosumab, glucocorticoids, or potassium supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in super saturation of calcium oxalate | 4-6 weeks
  Change in urine calcium oxalate supersaturation from baseline to the final follow-up visit, measured via 24-hour urine collection. This is a marker that can be predictive of stone episodes, as recurrent stones may take years to develop.

SECONDARY OUTCOMES:
Changes in urinary oxalate levels | 4-6 weeks
  Difference in 24-hour urinary oxalate excretion from baseline to the final follow-up visit, measured in mg/day, to assess the effect of dietary and pharmacologic interventions on oxalate levels.
Changes in urinary calcium levels | 4-6 weeks
  Difference in 24-hour urinary calcium excretion from baseline to the final follow-up visit, measured in mg/day, to evaluate the effect of chlorthalidone and dietary interventions on urinary calcium levels.
Chlorthalidone Adherence Survey (adapted from Brief Medication Questionnaire) | 4-6 weeks
  Participant-reported adherence to prescribed chlorthalidone therapy, assessed via a structured survey at the follow-up visit, to evaluate compliance with the study intervention.
  Response will be either 0=nonadherent or 1=adherent.

CONTACTS AND LOCATIONS:
Overall Officials: Mantu Gupta, MD, Principal Investigator — Mount Sinai West
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because all results are part of standard clinical care, and participants have access to their own medical records.